CLINICAL TRIAL: NCT00374673
Title: Efficacy of Repetitive Transcranial Magnetic Stimulation in the Treatment of Chronic Idiopathic Pain Syndromes : a Double Blind Sham Controlled Study
Brief Title: Efficacy of Transcranial Magnetic Stimulation (TMS) in Chronic Idiopathic Pain Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Nadine ATTAL, Clinical principal investigator, Hospital Ambroise Paré Paris
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMS-chronic pain 1
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Fibromyalgia; Irritable Bowel Syndrome; Burning Mouth Syndrome
Keywords: TMS; chronic pain; fibromyalgia; IBS; burning mouth syndrome; predictive factors
MeSH Terms: conditions — Fibromyalgia; Irritable Bowel Syndrome; Burning Mouth Syndrome; Chronic Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- transcranial magnetic stimulation (Experimental): repetitive transcranial magnetic stimulation of the motor cortex
  Interventions: Device: Repetitive transcranial magnetic stimulation
- placebo stimulation (Sham Comparator): repetitive placebo stimulation of the motor cortex
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation of the motor cortex (10 Hz) every day during 5 days then every week for 3 weeks then every two weeks for 2 months then every month for 3 additional months
  Other Names: placebo stimulation; rTMS

SUMMARY:
Objectives : To investigate the analgesic effects of repeated sessions of unilateral rTMS in patients with chronic pain syndrome due to fibromyalgia, IBS or burning mouth syndrome. Primary outcome will be numerical pain scores.

Methods : The study will be randomized and performed in parallel groups and double blind versus sham stimulation, and will include 90 patients (45 patients per treatment arm). The randomization will be computerized and performed for each aetiological group separately. The rTMS will be performed on the left motor cortex, 5 consecutive days , then once a week during 3 weeks then twice a month during 2 months, then once a month during 6 months. Clinical assessment will include an assessment of pain, quality of life, sleep, depression and anxiety, catastrophizing, and a neuropsychological evaluation.

Conclusion : this study should allow to determine for the first time the long term efficacy and safety of rTMS in the treatment of dysfunctional or idiopathic chronic pain syndromes which are often refractory to conventional treatments.

DETAILED DESCRIPTION:
Several lines of evidence suggest that fibromyalgia syndrome, Irritable Bowel syndrome (IBS) and burning mouth syndrome are chronic pain disorders affecting pain modulation. Repetitive transcranial magnetic stimulation (rTMS) is a recent, safe and non-invasive technique for stimulating the cerebral cortex, which has recently been reported to induce short term analgesic effects in patients with chronic focal pain. We have also recently shown in a double blind randomized trial, that rTMS could have short term analgesic effects in patients with fibromyalgia.

Objectives : Our aim is to investigate the long term analgesic effects of repeated sessions of unilateral rTMS in patients with chronic pain syndrome due to fibromyalgia, IBS or burning mouth syndrome. Primary outcome will be numerical pain scores on brief pain inventory at each visit.

Methods : This study will be randomized and performed in parallel groups and double blind versus sham stimulation. It will include at least 30 patients per pain disorder, ie 90 patients. Randomization will be computerized and performed for each of the aetiological groups separately (ie, there will be 3 distinct randomization procedures for fibromyalgia, IBS and stomatodynia);. Stimulation will be applied to the right motor area corresponding to the contralateral hand. The treatment will consist in a first period of 5 consecutive days of stimulation, followed by a stimulation once a week during 3 weeks then a stimulation twice a month during 2 months then stimulation once a month during 3 additional months. Clinical assessment will be performed at baseline, then at day 1, 5, weeks 3, 5, 7, 9, 13 and 25. It will include depending on the visits an assessment of pain intensity and characteristics, quality of life, sleep, depression and anxiety, catastrophizing, and a brief neuropsychological evaluation (focusing on memory, attention and vigilance). In patients with fibromyalgia, the evaluation will also include specifically the number of tender points. In patients with IBS, evaluation of bowel dysfunction will also be performed.

Conclusion : This study should allow to determine for the first time the long term efficacy and safety of rTMS in the treatment of dysfunctional or idiopathic chronic pain syndromes which are often refractory to conventional treatments.

ELIGIBILITY:
Inclusion Criteria:

* Pain related to Fibromyalgia (ACR criteria) or IBS (Rome II criteria) or burning mouth syndrome (IHS criteria 2004)
* Chronic pain for at least 6 months
* Pain for at least 4 days a week
* Mean average pain score at inclusion and randomization ≥ 4/10 (numerical scale)
* Patients aged 18 years and less than 80 years
* Informed consent
* Stable antalgic treatment

Exclusion Criteria:

* Contraindications to TMS (electroconvulsive therapy, epilepsy, head trauma, intracranial hypertension, metallic clip, pace maker, pregnancy)
* Major depression (DSM IV criteria) or psychosis
* Disorder preventing an accurate understanding of the testing and protocol
* Intermittent pain
* Pain for less than 6 months
* Other pain more severe than the pain evaluated for the trial
* Alcohol/psychoactive drugs abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-10; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Average pain over the last 24 hours at each visit -pain diary at baseline to see the stability of the measures | at each visit before the stimulation session
  Brief Pain inventory

SECONDARY OUTCOMES:
Sensory and affective pain scores (McGill pain questionnaire) | at baseline, then day 1, 5, weeks 3, 9, and 25 after the induction phase
  Short form MPQ was used
Quality of life (brief pain inventory) | at baseline, days 1, 5,weeks 3, 9, and 25 after the induction phase
  Brief Pain inventory (Cleeland and Ryan 1992) interference items (7)
Disability ( FIQ) | at days 1, 5, weeks 3, 9 and 25 after the induction phase
  FIQ only for fibromyalgia patients
Comorbidities (HAD) | at week 3 7, 13, 25 after the induction phase
  21 item Hospital anxiety and depression scale
Catastrophizing (PCS) | at weeks 3, 7, 13 and 25 after the induction phase
  Pain Catastrophizing Scale (Sullivan et al 1995)
Predictors of the response based on psychological factors and measures of cortical excitability | at inclusion
Safety including cognitive evaluation | at 6 months (cognitive evaluation) ; safety assessed every month for up to 12 months
  Cognitive tests were performed by a neuropsychologists and included measures of attention and memory
Comparison of the efficacy of TMS between 3 different pain disorders | during the whole study period -ie, days 1, 5, then before each stimulation throughout the study
  this can only be made when the two other groups of patients will have finished the enrollment - for now the study on fibromyalgia is finished and results analysed - the other groups are still being recruited (ie, IBS, burning mouth syndrome)
assessment of cortical excitability | day 1, 5, weeks 3, 9 and 21 after the induction phase
  determination of rest motor threshold, suprathreshold motor evoiked potentials (MEP), SICI and ICF, for the left hemisphere

CONTACTS AND LOCATIONS:
Overall Officials: Nadine ATTAL, MD, PhD, Principal Investigator — INSERM U 987 and AP-HP
Locations (1):
- Hôpital Ambroise Paré, Boulogne, France